CLINICAL TRIAL: NCT04487782
Title: Pragmatic Weight Loss Intervention During Menopause
Acronym: WISE
Status: Completed | Type: Observational
Sponsor: Kara Marlatt (Other)
Responsible Party: Sponsor-Investigator, Kara Marlatt, Assistant Professor-Research, Pennington Biomedical Research Center
Organization: Pennington Biomedical Research Center (Other)
Other Study IDs: PBRC 2019-056
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Menopause; Menopause Related Conditions
MeSH Terms: interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- High SES / African-American Women: Semi-structured focus groups of 6 to 8 women per group will be conducted. Women in these groups will be of higher socioeconomic status (SES) and will be African-American/Black.
  Interventions: Other: Focus Groups
- High SES / Caucasian Women: Semi-structured focus groups of 6 to 8 women per group will be conducted. Women in these groups will be of higher socioeconomic status (SES) and will be Caucasian/White.
  Interventions: Other: Focus Groups
- Low SES / African-American Women: Semi-structured focus groups of 6 to 8 women per group will be conducted. Women in these groups will be of lower socioeconomic status (SES) and will be African-American/Black.
  Interventions: Other: Focus Groups
- Low SES / Caucasian Women: Semi-structured focus groups of 6 to 8 women per group will be conducted. Women in these groups will be of lower socioeconomic status (SES) and will be Caucasian/White.
  Interventions: Other: Focus Groups

INTERVENTIONS:
Other: Focus Groups — The investigators are enrolling up to 56 women (total) to participate in semi-structured focus groups of 6-8 women per group conducted either in-person or virtually (online) to help us tailor a lifestyle intervention for midlife women during perimenopause.

SUMMARY:
The investigators are using a community-based participatory research (CBPR) model to develop a lifestyle intervention targeting weight loss that is specifically tailored to women in perimenopause.

DETAILED DESCRIPTION:
This is a participatory research study which will enroll women (n of up to 56) with experience of menopause to help identify preferred strategies (modalities) for weight loss, which will combine calorie (dietary) restriction and exercise tactics.

Aim 1: Explore attitudes and perceptions about weight gain during the menopause transition, and identify weight loss strategies from the patient (peer) perspective.

- The investigators will apply these learnings: 1) to understand barriers for weight management during menopause; 2) to establish strategies to guide retention; 3) to finalize the intervention structure, including feedback on the frequency and duration of the study visits; and 4) to gather feedback on menopause-specific education resources set to be provided throughout the intervention.

Aim 2: Engage the Community Advisory Board (CAB) of the Louisiana Clinical and Translational Center (LA CaTS) to understand scalability and community-based implementation of an intervention tailored for women in perimenopause.

- The investigators will then utilize the Louisiana Clinical & Translational Science Center (LA CaTS) Community Advisory Board (CAB) to help us tailor a lifestyle intervention in perimenopausal women with emphasis on scalability and community-based implementation using learnings obtained from the focus groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 60 years
* Currently experiencing (or have experienced) the one of the following menopause-related traits:
* Vasomotor symptoms including hot flashes and/or night sweats
* Irregular menstrual cycle
* African-American (Black) or Caucasian (White) race
* Self-report having a desire to lose (or maintain) weight during menopause
* Willing to be recorded during the focus group for transcription purposes

Exclusion Criteria:

* Are pre-menopausal
* Non-English speaking

Ages: 45 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: The investigators will enroll up to 56 women who self-report having experience of menopause and a desire to lose (or maintain) weight during menopause. An equal distribution of African-American (AA) and Caucasian women stratified by socioeconomic status (SES) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Duration | 1 day
  Identify how long would women prefer the intervention to last (e.g., number of months).
Motivation | 1 day
  Identify what motivates women (e.g., group setting, incentives, etc.).
Time Commitment | 1 day
  Identify how many times (e.g., days per week) that women would want to participate in a lifestyle intervention.
Diet | 1 day
  Identify the types of diets (e.g., keto, Mediterranean, intermittent fasting, etc.) that women have attempted before, and which diets they liked best.
Exercise | 1 day
  Identify the types of exercises (e.g., swimming, walking, weight training, etc.) that women like to do or would like to try.
Location | 1 day
  Identify where women would want to go to receive a lifestyle intervention (e.g., at Pennington, in local fitness centers, virtual/online, etc.).
Barriers | 1 day
  Identify specific barriers that women would encounter if participating in a lifestyle intervention.
Menopause Education | 1 day
  Identify specific education topics that women would like to receive as part of their lifestyle intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Kara L Marlatt, PhD, MPH, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kracht CL, Romain JS, Hardee JC, Santoro N, Redman LM, Marlatt KL. "It just seems like people are talking about menopause, but nobody has a solution": A qualitative exploration of menopause experiences and preferences for weight management among Black women. Maturitas. 2022 Mar;157:16-26. doi: 10.1016/j.maturitas.2021.11.005. Epub 2021 Nov 7. PMID 35120668